CLINICAL TRIAL: NCT00319787
Title: A Randomized Placebo Controlled Study to Assess the Rate of PSA Decrease, Anatomical & Metabolic Changes in the Prostate Determined by MRI/3D-MRS & Histological Changes by Biopsy in Subjects With Locally Advanced Prostate Carcinoma Treated With Either Casodex® (Bicalutamide) Alone or the Combination of Casodex® & ZD1839 (Iressa™)
Brief Title: Combination Casodex® and Iressa™ in Locally Advanced Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1839IL/0129
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Locally Advanced Prostate Cancer
MeSH Terms: interventions — Gefitinib

INTERVENTIONS:
Drug: Iressa

SUMMARY:
The purpose of this study is to determine if the addition of ZD1839 Iressa™ to standard treatment with Casodex® (bicalutamide) for locally advanced prostate cancer can detect a difference in the rate of decrease of prostate specific antigen (PSA) levels.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age. Men with histologically confirmed locally advanced prostatic adenocarcinoma

Exclusion Criteria:

* No prior treatment for prostate cancer, including surgery, radiotherapy, cryotherapy or thermotherapy. No abnormal laboratory values. No co-existing malignancies and any other significant clinical disorder or laboratory finding.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102
Dates: Start 2003-12; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Determine the difference in the rate of PSA decrease between treatments over a 6 months period.

SECONDARY OUTCOMES:
To detect changes in prostatic metabolites by using in vivo magnetic resonance spectroscopy (MRS)
To detect changes in prostate gland using magnetic resonance imaging (MRI)
To detect changes in serum tumor markers
To assess histopathological changes

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Norway Medical Director, MD, Study Director — AstraZeneca AS
Locations (3):
- Norway (3):
  - Research Site, Moelv
  - Research Site, Oslo
  - Research Site, Trondheim